CLINICAL TRIAL: NCT00011570
Title: Electrical Control of Bladder in Spinal Cord Injury Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bodner, Donald - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1770R
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Spinal Cord Injury
Keywords: defecation; electrical stimulation; penile erection; Spinal cord injury; urology
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (1):
- 1 (Other)
  Interventions: Device: Bladder & Bowel Control

INTERVENTIONS:
Device: Bladder & Bowel Control

SUMMARY:
The investigators will continue their work with implanted stimulators to improve bladder and bowel function. Electrical stimulation produces simultaneous contraction of sphincters with the target organs, making emptying difficult. By optimizing electrode placement, employing a new electrode design and waveform choice, it is hoped to improve the 50% of subjects able to defecate with existing approaches. This is part of a multi-center study with multiple support sources, including Rehab R&D, PVA and a commercial stimulator company.

ELIGIBILITY:
Inclusion Criteria:

Spinal cord injury with bowel & bladder problems

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-04; Primary Completion 2005-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bodner, MD, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States